CLINICAL TRIAL: NCT05152693
Title: Effects of Variety and Portion Size on Meal Intake of Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study design has changed.
Sponsor: Penn State University (Other)
Collaborators: Jenny Craig, Inc. (Industry)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of The Laboratory For The Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FoodVariety101
Record Dates: First submitted 2021-11-17; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior | interventions — Beverages

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Low Variety Small Portion Without Beverage (Experimental): Test meal with food components mixed together (low variety) with a small portion of food served without water
  Interventions: Other: Low variety; Other: Small Portion Size; Other: Without Beverage
- High Variety Small Portion Without Beverage (Experimental): Test meal with food components separated on the plate (high variety) with a small portion of food served without water
  Interventions: Other: High Variety; Other: Small Portion Size; Other: Without Beverage
- Low Variety Small Portion With Beverage (Experimental): Test meal with food components mixed together (low variety) with a small portion of food and water
  Interventions: Other: Low variety; Other: Small Portion Size; Other: With Beverage
- High Variety Small Portion With Beverage (Experimental): Test meal with food components separated on the plate (high variety) with a small portion of food and water
  Interventions: Other: High Variety; Other: Small Portion Size; Other: With Beverage
- Low Variety Large Portion With Beverage (Experimental): Test meal with food components mixed together (low variety) with a large portion of food and water
  Interventions: Other: Low variety; Other: Large Portion Size; Other: With Beverage
- High Variety Large Portion With Beverage (Experimental): Test meal with food components separated on the plate (high variety) with a large portion of food and water
  Interventions: Other: High Variety; Other: Large Portion Size; Other: With Beverage

INTERVENTIONS:
Other: Low variety — Meal components are mixed together on the plate
  Arms: Low Variety Large Portion With Beverage; Low Variety Small Portion With Beverage; Low Variety Small Portion Without Beverage
Other: High Variety — Meal components are served separately on the plate
  Arms: High Variety Large Portion With Beverage; High Variety Small Portion With Beverage; High Variety Small Portion Without Beverage
Other: Small Portion Size — Small meal portion size
  Arms: High Variety Small Portion With Beverage; High Variety Small Portion Without Beverage; Low Variety Small Portion With Beverage; Low Variety Small Portion Without Beverage
Other: Large Portion Size — Large meal portion size
  Arms: High Variety Large Portion With Beverage; Low Variety Large Portion With Beverage
Other: With Beverage — Meal served with water
  Arms: High Variety Large Portion With Beverage; High Variety Small Portion With Beverage; Low Variety Large Portion With Beverage; Low Variety Small Portion With Beverage
Other: Without Beverage — Meal served without water
  Arms: High Variety Small Portion Without Beverage; Low Variety Small Portion Without Beverage

SUMMARY:
The primary purpose of this study is to gain a better understanding of the combined effects of meal variety and portion size on food intake at a meal. The study will also explore relationships with eating microstructure such as eating rate and bite size. Additionally, other individual characteristics will be examined for their influence on the effects of variety and portion size on meal intake.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to travel to Penn State University Park campus weekly for meals
* Be fully vaccinated against COVID-19
* Be a woman 20 - 65 years old
* Regularly eat 3 meals/day
* Be willing to refrain from drinking alcohol the day before and during test days
* Have a body mass index between 18.0 and 35.0 kg/m*m
* Be willing to refrain from eating after 10 pm the evening before test sessions
* Be willing to participate in all study procedures

Exclusion Criteria:

* Must not be a smoker
* Must not be an athlete in training
* Must not be pregnant or breastfeeding at the time of screening
* Must not have taken prescription or non-prescription drugs that may affect appetite or food intake within the last 3 months
* Must not dislike or be unable to eat the test foods (because of allergies, intolerance, or dietary restrictions)
* Must not be currently dieting to gain or lose weight
* Must not have a health condition that affects appetite
* Must not have participated in a similar study in our lab in the past year
* Must not be a student, faculty, or staff member in nutritional sciences or psychology

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-20 (Estimated); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-01-27 (Estimated)

PRIMARY OUTCOMES:
Change in intake by weight | Weeks 1, 2, 3, 4, 5, 6
  Weight (grams) of all meal components consumed
Change in energy intake | Weeks 1, 2, 3, 4, 5, 6
  Energy intake (kilocalories) of all meal components consumed, calculated from weight and energy density

SECONDARY OUTCOMES:
Change in bite count | Weeks 1, 2, 3, 4, 5, 6
  The number of bites of food during the meal
Change in meal duration | Weeks 1, 2, 3, 4, 5, 6
  Duration of the meal in minutes
Change in mean eating rate | Weeks 1, 2, 3, 4, 5, 6
  Mean food intake per minute (grams/minute), calculated by dividing meal food intake by meal duration
Change in mean bite size | Weeks 1, 2, 3, 4, 5, 6
  Mean food intake per bite (grams/bite), calculated by dividing meal food intake by bite count
Change in sip count | Weeks 1, 2, 3, 4, 5, 6
  The number of sips of water during the meal
Change in mean drinking rate | Weeks 1, 2, 3, 4, 5, 6
  Mean water intake per minute (grams/minute), calculated by dividing meal water intake by meal duration
Change in mean sip size | Weeks 1, 2, 3, 4, 5, 6
  Mean water intake per sip (grams/sip), calculated by dividing meal water intake by sip count
Change in switching between bites and sips | Weeks 1, 2, 3, 4, 5, 6
  The number of switches between bites and sips during the meal
Change in rating of pleasantness of the taste of food samples | From before the test meal to after the test meal in weeks 1, 2, 3, 4, 5, 6
  Measured on a 100-mm visual analogue scale ranging from not at all pleasant (0 mm) to extremely pleasant (100 mm). This will be used to calculate Sensory-Specific Satiety
Change in rating of prospective consumption of food samples | From before the test meal to after the test meal in weeks 1, 2, 3, 4, 5, 6
  Measured on a 100-mm visual analogue scale ranging from none at all (0 mm) to vary large amount (100 mm) how much of [this food] do you want to eat right now?. This will be used to calculate Sensory-Specific Satiety
Change in rating of hunger | From before the test meal to after the test meal in weeks 1, 2, 3, 4, 5, 6
  Measured on a 100-mm visual analogue scale ranging from not at all hungry (0 mm) to extremely hungry (100 mm)
Change in rating of thirst | From before the test meal to after the test meal in weeks 1, 2, 3, 4, 5, 6
  Measured on a 100-mm visual analogue scale ranging from not at all thirsty (0 mm) to extremely thirsty (100 mm)
Change in rating of nausea | From before the test meal to after the test meal in weeks 1, 2, 3, 4, 5, 6
  Measured on a 100-mm visual analogue scale ranging from not at all nauseated (0 mm) to extremely nauseated (100 mm)
Change in rating of fullness | From before the test meal to after the test meal in weeks 1, 2, 3, 4, 5, 6
  Measured on a 100-mm visual analogue scale ranging from not at all full (0 mm) to extremely full (100 mm)
Change in rating of prospective consumption of the meal | At the start of the test meal in weeks 1, 2, 3, 4, 5, 6
  Measured on a 100-mm visual analogue scale ranging from nothing at all (0 mm) to a large amount (100 mm) in answer to the question 'How much food could you eat right now?'.
Change in rating of the size of the meal compared to participant's usual portion | At the start of the test meal in weeks 1, 2, 3, 4, 5, 6
  100-point visual analog scale ranging from a lot smaller (0 mm) to a lot larger (100 mm)
Change in rating of how filling the participant expects this amount of food to be | At the start of the test meal in weeks 1, 2, 3, 4, 5, 6
  100-point visual analog scale ranging from not at all filling (0 mm) to extremely filling (100 mm)
Change in rating of meal termination due to fullness | At the end of the test meal in weeks 1, 2, 3, 4, 5, 6
  100-point visual analog scale ranging from strongly disagree (0 mm) to strongly agree (100 mm)
Change in rating of meal termination due to eating their usual amount | At the end of the test meal in weeks 1, 2, 3, 4, 5, 6
  100-point visual analog scale ranging from strongly disagree (0 mm) to strongly agree (100 mm)
Change in rating of meal termination due to eating is no longer a priority | At the end of the test meal in weeks 1, 2, 3, 4, 5, 6
  100-point visual analog scale ranging from strongly disagree (0 mm) to strongly agree (100 mm)
Change in rating of meal termination due to there being no food left | At the end of the test meal in weeks 1, 2, 3, 4, 5, 6
  100-point visual analog scale ranging from strongly disagree (0 mm) to strongly agree (100 mm)
Change in rating of meal termination due to self-consciousness about amount consumed | At the end of the test meal in weeks 1, 2, 3, 4, 5, 6
  100-point visual analog scale ranging from strongly disagree (0 mm) to strongly agree (100 mm)
Change in rating of meal termination due to the food no longer tasting good | At the end of the test meal in weeks 1, 2, 3, 4, 5, 6
  100-point visual analog scale ranging from strongly disagree (0 mm) to strongly agree (100 mm)
Change in estimation of proportion of meal eaten | At the end of the test meal in weeks 1, 2, 3, 4, 5, 6
  100-point visual analog scale ranging from 0% to 100%
Change in estimation of calories consumed at the meal | At the end of the test meal in weeks 1, 2, 3, 4, 5, 6
  Open ended question (number of calories)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for the Study of Human Ingestive Behavior, The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No